CLINICAL TRIAL: NCT06499246
Title: Parathyroid Allotransplant for Severe Refractory Hypoparathyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Devon (Other)
Collaborators: University Health Network, Toronto (Other); University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Karen Devon, Associate Professor of Surgery, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5129
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Hypoparathyroidism Postprocedural

STUDY DESIGN:
Intervention Model Description: Parathyroid transplant from brain dead donors into patients with permanent hypoparathyroidism
Masking Description: It is open label. No masking involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parathyroid Transplant (Experimental): Patients with permanent refractory hypoparathyroidism after total thyroidectomy will be entered in this study to undergo parathyroid transplantation from a neurologically deceased donor. Inclusion criteria are patients who have had a prior total thyroidectomy with both biochemical hypoparathyroidism and symptomatic hypocalcemia (numbness, tingling, or other neurologic symptoms) requiring daily high dose calcium (greater than 2000 mg per day), vitamin D (greater than 2 mcg of calcitriol per day) supplementation and/or intermittent IV calcium infusion. Patients for inclusion must have failed this medical management after at least 1 year of treatment and meet standard criteria for receiving organ transplant.
  Interventions: Procedure: Donor Parathyroid

INTERVENTIONS:
Procedure: Donor Parathyroid — Once a potential donor becomes available, the transplant team will assess if the donor is a match for our study participant using standardized transplantation protocols that include serology blood tests completed in the pre-operative setting. If the donor is a match, the procurement team will procure all parathyroid tissue using standard surgical techniques. The specimen will be kept in organ preservation solution for transport and transported to the operating room. The recipient (study participant) will be admitted to the hospital under and taken to the operating room for the surgical procedure. Once the procurement team arrives with the parathyroid tissue the procedure will be performed under local anesthesia using a well-established technique, for parathyroid auto transplant, of implanting parathyroid tissue in the non-dominant brachioradialis muscle. Immunosuppression medication protocols will be initiated.

SUMMARY:
Hypoparathyroidism following thyroid surgery presents significant challenges, often leading to debilitating symptoms and reduced quality of life despite conventional treatment. Having now reported the first successful case of a deceased donor fresh tissue parathyroid allotransplant with immunosuppression in a transplant-naive recipient, the purpose of this study is to further assess the safety and efficacy of this procedure in patients with severe intractable post-surgical hypoparathyroidism.

DETAILED DESCRIPTION:
A protocol for deceased donor parathyroid transplantation was developed with the University Health Network Ajmera Transplant Centre in Toronto, relevant stakeholders, and presented to the innovation committee and REB for approval. Health Canada approval was obtained under the scope of existing cell tissue and organ regulations within the provincial organ procurement agency.

This is a pilot, prospective case-series. It includes a cohort of patients with hypoparathyroidism who will undergo parathyroid transplantation from a neurologically deceased donor. There is no control group in this study.

Patients with permanent refractory hypoparathyroidism after total thyroidectomy will be entered in this study to undergo parathyroid transplantation from a neurologically deceased donor. Inclusion criteria are patients who have had a prior total thyroidectomy with both biochemical hypoparathyroidism and symptomatic hypocalcemia (numbness, tingling, or other neurologic symptoms) requiring daily high dose calcium (greater than 2000 mg per day), vitamin D (greater than 2 mcg of calcitriol per day) supplementation and/or intermittent IV calcium infusion. Patients for inclusion must have failed this medical management after at least 1 year of treatment and meet standard criteria for receiving organ transplant.

All patients will have at least one pre-operative clinic visit with the endocrine surgery, endocrinology, and transplant team for comprehensive assessment. Baseline blood work will be conducted at this pre-operative visit, as outlined in the study protocol. The patient will also be evaluated by psychiatry and complete any necessary age appropriate comprehensive cancer screening as per standard transplantation protocol. Completeness of pre-transplant vaccinations (pneumococcus, HBV, influenza, Tdap, HAV) will be reviewed and arranged in co-ordination with patients' primary care provider as necessary. If based on pre-transplant work up a participant is deemed to meet exclusion criteria and not be suitable for transplant this will be discussed with the participant, and they will be withdrawn from the study. Participants will be informed of the need to fulfill the previously listed standard transplant criteria during the informed consent process.

Once a potential donor becomes available, the transplant team will decide whether the donor is a match for a study participant. A rigorous protocol for donor selection and transplantation was developed. Donor criteria aimed at minimizing infectious and immunological risks (HLA matching). A history of hyperparathyroidism (primary, secondary or tertiary) will also be screened for in the donor as the presence of hyperparathyroidism would be an exclusion criteria to procure their parathyroid glands for this study. If the donor is a match for a study participant, the participant will be contacted and timing of retrieval and patient arrival at TGH will be coordinated. The procurement team will then, with appropriate timing, procure all parathyroid tissue using standard surgical techniques and the tissue will be kept in organ preservation solution in a sterile specimen cup with a cold ischemic time of less than 2 hours.

The study participant will be admitted to the hospital under the Multi Organ Transplant team at TGH and will be taken to the operating room for the surgical procedure. The procedure will be performed under local anesthesia using a well-defined technique in the non-dominant brachioradialis muscle. The length of the surgery is estimated to be less than an hour. The patient will be recovering in PACU and then transferred back to the ward after the procedure is completed for continuation of the immunosuppressive therapy according to an established UHN Multiorgan Transplant protocol. After monitoring overnight, the patient will be discharged home the day following surgery.

The patient will be discharged home on day 1 post surgery and follow up will be arranged on day 3 and day 7 in for monitoring of calcium profile and response to treatment. Long-term follow-up for the patient will occur at 1, 3 and 12 months post-operatively with the endocrine surgery, endocrinology and transplant teams.

The primary outcomes of the study are to assess improvement in hypoparathyroidism as assessed by biochemistry and patient symptoms with secondary outcomes including risk of surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Prior total thyroidectomy
* Symptomatic hypocalcemia (numbness, tingling, or other neurologic symptoms) requiring daily high dose calcium (greater than 2000 mg per day) and vitamin D (greater than 2 mcg of calcitriol per day) supplementation and/or intermittent IV calcium infusion.
* Biochemical blood test consistent with hypoparathyroidism
* Failed medical management (>1 year of post-thyroidectomy hypoparathyroidism treated medically with persistent biochemical disease and symptoms)
* Patient meets current standards for receiving an organ transplant (e.g. no active infection, no malignancy, no contraindications to immunosuppression or surgery)

Exclusion Criteria:

* <18 years old male or female
* Current pregnancy
* Advanced stage 3-4 thyroid cancer
* Contraindication to surgery or immunosuppression
* Malignancy with contraindication to transplant:

  1. Certain active malignancies are not a contraindication to transplant such as prostate cancer or lymphoproliferative disease in remission, and locoregional skin malignancies such as melanoma will be transplant candidates (outlined in Preexisting melanoma and hematological malignancies, prognosis, and timing to solid organ transplantation: A consensus expert opinion statement by Al-Adra et al respectively).
  2. Remote malignancies with successful treatment will not preclude patients from inclusion in the study. Dependent upon the malignancy risk level a minimal time from treatment will be required as established by the consensus recommendations outlined in Pretransplant solid organ malignancy and organ transplant candidacy: A consensus expert opinion statement by Al-Adra et al.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Maintain calcium levels without standard calcium replacement treatment. | Pre-operatively and then at 4 weeks, 3 months and 12 months post-operatively
  Patients will demonstrate improvement in hypocalcemia symptoms, biochemical calcium profile, and parathyroid hormone levels as well as decrease frequency of emergency visits for intravenous calcium. Specifically at each assessment patients will be questioned regarding numbness and tingling and will be examined for presence of Chvostek's and Trousseau's sign. Additionally, to assess overall impact of symptoms in relation to quality of life. A hypoparathyroidism quality-of-life questionnaire will be filled out by the patient pre-operatively and at 12 months post-operatively. This questionnaire was formulated and has been used for research purposes by the HypoParaUK group. Biochemical calcium profile (serum total calcium, albumin, ionized calcium, parathyroid hormone level, vitamin D level, phosphate) using blood tests done on post-operative day 1, 3, 5, 7, and subsequently 2 weeks, 3 weeks, 4 weeks post-operatively, and afterwards monthly for a total of 12 months post-operatively.

SECONDARY OUTCOMES:
Rate of surgical complications | 4 weeks, 3 months and 12 months post-operatively
  Whether parathyroid allotransplant from neurologically deceased donors amongst patients with permanent refractory hypoparathyroidism has minimal surgical and medical complications and the need for medications.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Devon, MD, MSc, FRCSC, FACS, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kim E, Ramonell KM, Mayfield N, Lindeman B. Parathyroid allotransplantation for the treatment of permanent hypoparathyroidism: A systematic review. Am J Surg. 2022 Apr;223(4):652-661. doi: 10.1016/j.amjsurg.2021.07.025. Epub 2021 Jul 20. PMID 34304848
- [Background] Devon K, Tinckam K, Humar A, Madani A, Pasternak JD, Saravana-Bawan B, Zahedi A. Successful Deceased Donor Parathyroid Allotransplantation: A Novel Approach in a Patient with Severe Refractory Hypoparathyroidism After Thyroidectomy for Thyroid Cancer. Thyroid. 2024 Aug;34(8):1058-1061. doi: 10.1089/thy.2024.0115. Epub 2024 Jul 18. No abstract available. PMID 38919120